CLINICAL TRIAL: NCT02992210
Title: Multicenter Trial of Phase I/II Studies on GD2 Positive Solid Tumors by 4SCAR-GD2
Brief Title: Study on GD2 Positive Solid Tumors by 4SCAR-GD2
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Principal Investigator, Lung-Ji Chang, Director, Shenzhen Geno-Immune Medical Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-16002
Record Dates: First submitted 2016-12-03; First posted 2016-12-14 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor
Keywords: CAR; chimeric antigen receptor; adoptive T cell transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- effectiveness of 4SCAR-GD2 T cells (Experimental): The 4SCAR-GD2-modified T cells can recognize and kill tumor cells through the recognize of GD2 .This study will evaluate the side effects and effective doses of 4SCAR-GD2 T cells in treating refractory and recurrent solid tumors
  Interventions: Genetic: 4SCAR-GD2

INTERVENTIONS:
Genetic: 4SCAR-GD2 — GD2-specific 4th Generation CART
  Other Names: GD2-specific 4th Generation CART

SUMMARY:
Patients with refractory and/or recurrent solid tumor have poor prognosis despite complex multimodel therapy and therefore, novel approaches are urgently needed. The investigators are attempt to treat these diseases using T cells genetically modified with a 4th generation lentiviral chimeric antigen receptor (4SCAR fused with an inducible apoptotic caspase 9 domain) targeting GD2 (4SCAR-GD2). The 4SCAR-GD2-modified T cells can recognize and kill tumor cells through the recognition of GD2, a surface protein expressed at high levels on many types of tumors but not on normal tissues. This study will evaluate the side effects and effective doses of 4SCAR-GD2 T cells in treating refractory and/or recurrent tumors.

DETAILED DESCRIPTION:
Background:

Patients with refractory and/or recurrent solid tumors have poor prognosis despite complex multimodal therapy; therefore, novel curative approaches are needed. The investigators are attempting to use T cells obtained directly from the patient, which can be genetically modified to express a 4th generation GD2-specific chimeric antigen receptor (4SCAR-GD2). The chimeric antigen receptor (CAR) molecules enable the T cells to recognize and kill tumor cells through the recognition of a surface antigen, GD2, which is expressed at high levels on tumor cells but not at significant levels on normal tissues. This study will evaluate the side effects and the best dose of a novel 4th generation anti-GD2 CAR T cells to refractory and/or recurrent solid tumors.

Design:

Participants will be screened through physical exam and medical history. Blood and urine samples will be collected. Imaging studies or bone marrow aspirates may be performed.

Peripheral blood mononuclear cells (PBMC) will be obtained by apheresis, and T cells will be activated and modified to express the 4SCAR-GD2 gene.

On Day -5 to -7, PBMC will be activated and enriched for T cells, which will be followed by 4SCAR-GD2 lentiviral transduction. The total culture time is approximately 5-7 days.

Participants will receive a preparative conditioning regimen comprising cyclophosphamide/fludarabine to prepare their immune system to accept the modified CAR T cells.The preparative regimen will be based on patient immune condition and consistent with standard chemotherapy conditioning regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients with tumors have received standard first-line therapy and been judged to be non-resectable，metastatic,progressive or recurrent.
* The GD2 antigen status of the tumor will be determined for eligibility.Positive expression is defined by GD2 antibody staining results based on immunohistochemistry or flow cytometry analyses.
* Body weight greater than or equal to 10 kg.
* Age: ≥1 year and ≤ 65 years of age at the time of enrollment.
* Life expectancy: at least 8 weeks.
* Prior Therapy: 1) There is no limit to the number of prior treatment regimens. Any grade 3 or 4 non-hematologic toxicity of any previous therapy must have resolved to grade 2 or less. 2) Must not have received hematopoietic growth factors for at least 1 week prior to mononuclear cells collection. 3) At least 7 days must have elapsed since the completion of therapy with a biologic agent, targeted agent, tyrosine kinase inhibitor or a metronomic nonmyelosuppressive regimen. 4) At least 4 weeks must have elapsed since prior therapy that included a monoclonal antibody. 5) At least 1 weeks since any radiation therapy at the time of study entry.
* Karnofsky/jansky score of 60% or greater.
* Cardiac function: Left ventricular ejection fraction greater than or equal to 40/55 percent .
* Pulse Ox greater than or equal to 90% on room air.
* Liver function: defined as alanine transaminase (ALT) <3x upper limit of normal (ULN), aspartate aminotransferase (AST) <3x ULN; serum bilirubin and alkaline phosphatase <2x ULN.
* Renal function: Patients must have serum creatinine less than 3 times upper limit of normal.
* Marrow function: White blood cell count ≥1000/ul, Absolute neutrophil count ≥500/ul, Absolute lymphocyte count ≥500/ul, Platelet count ≥25,000/ul (not achieved by transfusion).
* Patients with known bone marrow metastatic disease will be eligible for study as long as they meet hematologic function criteria, and the marrow disease not evaluable for hematologic toxicity.
* For all patients enrolled in this study, their parents or legal guardians must sign an informed consent and assent.

Exclusion Criteria:

* Existing severe illness (e.g. significant cardiac, pulmonary, hepatic diseases, etc.) or major organ dysfunction, with the exception of grade 3 hematologic toxicity.
* Untreated central nervous system (CNS) metastasis: Patients with previous CNS tumor involvement that has been treated and is stable for at least 6 weeks following completion of therapy are eligible.
* Previous treatment with other genetically engineered GD2-CAR T cells.
* Active HIV, Hepatitis B virus (HBV), Hepatitis C virus (HCV) infection or uncontrolled infection.
* Patients who require systemic corticosteroid or other immunosuppressive therapy.
* Evidence of tumor potentially causing airway obstruction.
* Inability to comply with protocol requirements.
* Insufficient CAR T cells availability.

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events. | 3 year
  Determine the toxicity profile the 4SCAR-GD2-modified T cells with Common Toxicity Criteria for Adverse Effects version 4.0

SECONDARY OUTCOMES:
Anti-tumor effects | 3 year
  Disease status is defined by the biochemical markers and image scan to get the outcomes such as Complete response/remission (CR) , Very good partial response/remission (VGPR) , etc
The expansion and persistence of anti-GD2 CAR T cells | 3 year
  The investigators will monitor the expansion and functional persistence of 4SCAR-GD2 T cells in the peripheral blood of patients and the correlation with antitumor effects
Immune responses after anti-GD2 infusions | 1 year
  assessment of lymphocyte phenotypes and anti-tumor activity
Immune responses after anti-GD2 infusions | 1 year
  assessment of cytokine profile
Survival time of the patients | 3 year
  Evaluate the survival time of the patients treated with the 4SCAR-GD2 T cells, including progression free survival (PFS) and overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, Principal Investigator — Shenzhen Geno-Immune Medical Institute
Locations (1):
- Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong, China